CLINICAL TRIAL: NCT04565028
Title: Functional Outcomes of Cannabis Use (FOCUS) in Veterans With Posttraumatic Stress Disorder
Acronym: FOCUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: D3276-R
Record Dates: First submitted 2020-09-18; First posted 2020-09-25 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: PTSD; Cannabis-Related Disorder
Keywords: PTSD; Cannabis-Related Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Marijuana Abuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Contingency Management (CM) (Experimental): Mobile contingency management (CM) will be used to promote reductions in cannabis use among Veterans with PTSD who are heavy cannabis users. CM is an intensive behavioral therapy in which participants are paid to reduce substance use.
  Interventions: Behavioral: Contingency Management (CM)

INTERVENTIONS:
Behavioral: Contingency Management (CM) — Contingency management is an intensive behavioral therapy in which participants are paid to reduce substance use.
  Other Names: Mobile Contingency Management (mCM)

SUMMARY:
Posttraumatic stress disorder (PTSD) is a disabling psychiatric disorder that affects 20%-30% of U.S. Veterans. PTSD is strongly associated with increased risk for substance abuse comorbidity, including cannabis use disorder. Multiple states now include PTSD as a condition for which patients can be legally prescribed medical marijuana, despite the fact that there has not been a single large-scale randomized clinical trial demonstrating the efficacy of cannabis to treat PTSD to date. The overall objective of the current proposal is to study the impact of reduced cannabis use on functioning among Veterans with PTSD. The investigators will evaluate the relationship between cannabis use and daily functioning among cannabis users and heavy cannabis users. The central hypothesis is that reductions in cannabis use will lead to positive changes in the functional outcomes of Veterans. The rationale for this research is that it will provide the first and only real-time data concerning the impact of reduced cannabis use on daily functioning among Veterans with PTSD.

DETAILED DESCRIPTION:
Posttraumatic stress disorder (PTSD) is a disabling psychiatric disorder that affects 20%-30% of U.S. Veterans. PTSD is strongly associated with increased risk for substance abuse comorbidity, including cannabis use disorder; however, multiple states now include PTSD as a condition for which patients can be legally prescribed medical marijuana, despite the fact that there has not been a single large-scale randomized clinical trial demonstrating the efficacy of cannabis to treat PTSD to date. The overall objective of the current proposal is to prospectively study the impact of reduced cannabis use on psychosocial functioning among Veterans with PTSD. To do so, the investigators will first use ecological momentary assessment (EMA) methods to evaluate the relationship between cannabis use and daily functioning among Veterans with PTSD. Next, the investigators will use mobile contingency management (CM) and EMA to assess the impact of reduced cannabis use on daily functioning among Veterans with PTSD who are heavy cannabis users. The central hypothesis is that reductions in cannabis use will lead to positive changes in the functional outcomes of Veterans. The rationale for this research is that it will provide the first and only real-time data concerning the impact of reduced cannabis use on daily functioning among Veterans with PTSD. As a result, this innovative and timely project has the potential to significantly advance VHA healthcare and will directly inform the ongoing national debate concerning the impact of cannabis use on the long-term functional recovery of Veterans with PTSD.

ELIGIBILITY:
Inclusion Criteria:

* Veteran status
* Ability to speak and write fluent English
* Current PTSD diagnosis
* Use of cannabis on 13+ days in the past month (i.e., use on 3+ days per week)

Exclusion Criteria:

Participants will be excluded if they:

* Have experienced a change in their psychiatric medication regimen during the past month (e.g., a new medication has been prescribed or the dose of an existing medication has been changed), or expect to experience a such a change during the course of the study
* Are receiving non-study CUD treatment
* Meet diagnostic criteria for bipolar disorder or schizophrenia (note that the SCID-5 (First et al., 2015) will be used to diagnoses these and other disorders)
* Become imprisoned
* Become hospitalized for psychiatric reasons
* Report imminent risk for suicide or homicide
* Meet current criteria for a substance use disorder other than cannabis use disorder or tobacco

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-01-26 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in functional impairment as measured by the World Health Organization Disability Assessment Schedule 2.0 (WHO-DAS) | Baseline and post-treatment (approximately six weeks)
  Functional impairment will be measured by the simple score on the World Health Organization Disability Assessment Schedule 2.0 (WHO-DAS). This measure has a scoring range of 0 to 144, with lower scores indicating lower functional impairment.
Change in functional impairment as measured by the Inventory of Psychosocial Functioning (IPF) | Baseline and post-treatment (approximately six weeks)
  Functional impairment will be measured by the Inventory of Psychosocial Functioning (IPF). This measure has a scoring range of 0 to 480, with lower scores indicating higher functional impairment.
Change in psychiatric distress | Baseline and post-treatment (approximately six weeks)
  Psychiatric distress will be measured by the 90-item Symptom Checklist (SCL-90). This measure has a scoring range of 0 to 360, with lower scores indicating lower distress related to mental health.
Change in quality of life, as measured by the WHOQOL-BREF | Baseline and post-treatment (approximately six weeks)
  Quality of life will be measured with the World Health Organization Quality of Life Brief (WHOQOL-BREF). The measure has a scoring range of 0 to 100, with higher scores denoting a higher quality of life.
Change in quality of life, as measured by the Quality of Life Scale | Baseline and post-treatment (approximately six weeks)
  Quality of life will be measured with the 16-item Quality of Life Scale. The measure has a scoring range of 6 to 112, with higher scores denoting a higher quality of life.
Change in number of days of drugged driving as measured by timeline follow-back | Baseline and post-treatment (approximately six weeks)
  Number of days of drugged driving in the past month will be self-reported by participants using a Timeline Follow-Back Interview.
Change in cannabis use | Baseline and post-treatment (approximately six weeks)
  Cannabis use, as measured in milligrams, will be measured by taking the product of number of days used and amount used per day in the previous week.

CONTACTS AND LOCATIONS:
Overall Officials: Jean C Beckham, PhD, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
The investigators do not plan to attend individual participant data.